CLINICAL TRIAL: NCT05166915
Title: Respiratory Application of a Novel Ultraviolet Light Delivery Device for Patients Infected With COVID-19: A Randomized, Sham-Controlled Study
Brief Title: Respiratory COVID-19: A Randomized, Sham-Controlled Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Indefinite hold by Company.
Sponsor: Aytu BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: UVL-0001
Record Dates: First submitted 2021-12-20; First posted 2021-12-22 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: COVID-19 Pneumonia; Acute Respiratory Distress Syndrome; COVID-19 Acute Respiratory Distress Syndrome; COVID-19 Respiratory Infection
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to receive treatment with the functional UVA light catheter or the sham control device.
Who Masked: Participant, Care Provider
Masking Description: Randomized, Sham Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- UVA Light Emitting Catheter (Experimental): Experimental Device intended to eliminate microorganisms using UV-A light, thereby reducing the viral burden of SARS-CoV-2.
  Interventions: Device: UVA Light Emitting Catheter
- Sham Control Device (Sham Comparator): Sham Control Device
  Interventions: Device: Sham Control Catheter

INTERVENTIONS:
Device: UVA Light Emitting Catheter — Experimental Device intended to eliminate microorganisms using UV-A light, thereby reducing the viral burden of SARS-CoV-2
  Arms: UVA Light Emitting Catheter
Device: Sham Control Catheter — Sham Control Device
  Arms: Sham Control Device

SUMMARY:
A study of intubated critically ill patients infected with SARS-COV-2 to evaluate the safety and treatment effects of ultraviolet-A (UVA) light administered by a novel device via endotracheal tube in a first-in-human study. Study hypothesis was that respiratory SARS-CoV-2 viral burden would significantly decrease following five (5) days of UVA therapy.

DETAILED DESCRIPTION:
The UV Respiratory Tract Light Therapy Device is intended to emit energy in the UVA region of the spectrum in intubated patients to reduce the viral burden of SARS-CoV-2 (human pathogenic coronavirus (COVID-19)) in intubated patients. The System is to be used in conjunction with the current standard of care measures.

The UV Respiratory Tract Light Therapy Device is intended to be used for 20 minutes per 24-hour period for the endotracheal application for 5 days, in combination with pharmacological and/or physical measures to optimize the therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age
2. Confirmed positive test result for SARS-CoV-2 within 14d
3. Mechanically ventilated (first intubation since positive SARS-CoV-2 test)
4. Endotracheal tube inner diameter at least 7.5 mm

Exclusion Criteria:

1. Unable to provide informed consent (or surrogate)
2. Enrolled in a therapeutic clinical trial for COVID-19 that does not allow recruitment in other trials.
3. Pregnant women. While not an exclusion criterion, special care should be exercised in treating patients who are receiving concomitant therapy (either topically or systemically) with known photosensitizing agents such as anthralin, coal tar or coal tar derivatives, griseofulvin, phenothiazines, nalidixic acid, fluoroquinolone antibiotics, halogenated salicylanilides (bacteriostatic soaps), sulfonamides, tetracyclines, thiazides and certain organic staining dyes such as methylene blue, toluidine blue, rose bengal, and methyl orange.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in viral load in endotracheal tube aspirates | Day 0-Day 5
  Difference in change in viral load from the endotracheal tube (ETT) aspirates on day 0 to the last day of treatment between treated and untreated subjects.

SECONDARY OUTCOMES:
Overall reduction or change of endotracheal bacterial content in upper airway | Day 0-Day 5
  Change in endotracheal bacterial content (determined by culture or PCR methodology) from the ETT aspirate on day 0 to the last day of treatment.
Days to extubation | Day 0 - Day 30
  Days to extubation
Development of ventilated associated pneumonia (VAP) | Day 0-Day7
  Percentage of development of VAP in between day 0 to day 7. VAP is defined by new or progressive pulmonary infiltrates on imaging along with clinical suspicion by the managing team (e.g. fever, leukocytosis, increased procalcitonin) warranting initiation or change in antibiotic therapy.
Days to discharge from hospital | Day 0 - Day 30
  Days to discharge from hospital
Mean ordinal scale on day 15 | Day 14
  1. Death
  2. Hospitalized, on invasive mechanical ventilation with additional organ support, ECMO, pressors, RRT
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  7. Not hospitalized, limitation on activities and/or requiring home-oxygen;
  8. Not hospitalized, no limitations on activities
Mean ordinal scale on day 28 | Day 27
  1. Death
  2. Hospitalized, on invasive mechanical ventilation with additional organ support, ECMO, pressors, RRT
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care;
  7. Not hospitalized, limitation on activities and/or requiring home-oxygen;
  8. Not hospitalized, no limitations on activities
Changes in Ferritin levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in Ferritin levels (4.63-204.0 ng/mL) day 0-7
Change in Interleukin-6 (IL-6) levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in interleukin-6 levels (Critical value: ≥ 100 pg/mL) day 0-7
Changes in C reactive protein levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in C reactive protein levels (<5 mg/L) day 0-7
Changes in White blood cell levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in White blood cell levels (4.00-11.00 x 1000/UL) day 0-7
Changes in Procalcitonin levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in Procalcitonin levels (<0.08 ng/mL) day 0-7
Changes in Lymphocyte counts (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in Lymphocyte count (1.00-4.50 x 1000/UL) day 0-7
Changes in D-dimer levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in D-dimer levels (0.00-0.50 µg/mL) day 0-7
Changes in Creatine Phosphokinase levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in Creatine Phosphokinase levels (29-168 U/L) day 0-7
Changes in Troponin levels (Exploratory Measure those drawn for clinical care) | Day 0 - Day 7
  Changes in Troponin levels (<0.04 ng/mL) day 0-7
Overall reduction or change of SARS-CoV-2 serum viral load (Exploratory Measure) | Day 0 - Day 5
  Change in viral load for blood serum sample on day 0 through the last day of treatment (Day 0, Day 1, Day 2, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Torres, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clinic of Barcelona, Barcelona, Catalan
  - Vall d'Hebron University Hospital, Barcelona, Catalan

IPD SHARING:
Plan to Share IPD: No